CLINICAL TRIAL: NCT05827159
Title: Emergency Department-Initiated Medications for Alcohol Use Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kathryn Hawk, Associate Professor of Emergency Medicine and Epidemiology (Chronic Disease), Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000034359; 1R01AA030568-01 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: Emergency Department; Brief Intervention; Naltrexone; Gabapentin
MeSH Terms: conditions — Alcoholism; Emergencies | interventions — Naltrexone; Gabapentin

STUDY DESIGN:
Intervention Model Description: Study participants will be identified through targeted screening for DSM-5 criteria for moderate to severe AUD and the study inclusion/exclusion criteria. Therefore, the Screening component of the SBIRT intervention in the proposed RCT will be conducted before eligible ED patients who are interested in study participation are consented and randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBIRT (Experimental): Participants will receive the Brief Negotiation Interview (BNI) and Referral to Treatment. The BNI has four key components: (1) permission to discuss substance use, (2) feedback on the health consequences of ongoing substance use, including making a connection between the ED visit and substance use, (3) motivational enhancement, and (4) negotiation and advice.
  Interventions: Behavioral: Brief Negotiation Interview
- SBIRT+ED-MAUD (Experimental): Participants with receive BNI, Referral to Treatment, and MAUD. In the MAUD component, either XR-NTX or oral naltrexone will be provided, supplemented by ancillary treatment with gabapentin. Participants will receive their first doses of XR-NTX (injection) and gabapentin in the ED and will receive 7 days of gabapentin take-home doses. Those who prefer to initiate treatment in ED with oral naltrexone receive their first doses of naltrexone and gabapentin in the ED and receive 29-day take-home doses of naltrexone and 7 days of gabapentin.
  Interventions: Drug: Naltrexone Pill; Drug: Naltrexone Injection; Behavioral: Brief Negotiation Interview; Drug: Gabapentin Pill

INTERVENTIONS:
Drug: Naltrexone Pill — In the MAUD component, some participants will receive oral Naltrexone in the ED.
  Other Names: Oral naltrexone
  Arms: SBIRT+ED-MAUD
Drug: Naltrexone Injection — In the MAUD component, some participants will receive a dose of XR-NTX (injection) in the ED.
  Other Names: XR-NTX
  Arms: SBIRT+ED-MAUD
Behavioral: Brief Negotiation Interview — Brief Negotiation Interview (BNI) has four key components: (1) permission to discuss substance use, (2) feedback on the health consequences of ongoing substance use, including making a connection between the ED visit and substance use, (3) motivational enhancement, and (4) negotiation and advice.
  Other Names: BNI
Drug: Gabapentin Pill — In the MAUD component, ancillary treatment with gabapentin will be provided.
  Other Names: Oral gabapentin
  Arms: SBIRT+ED-MAUD

SUMMARY:
The proposed study will be the first randomized clinical trial to evaluate a comprehensive Emergency Department (ED)-based intervention for moderate to severe Alcohol Use Disorder (AUD) combining Screening, Brief Intervention and Referral to Treatment (SBIRT) with ED-initiated medications for treatment of alcohol use disorder (MAUD).

The primary objective of this phase 3 study is to evaluate for differences in treatment engagement 30 days after ED visit between emergency department patients with moderate to severe alcohol use disorder (AUD) who are randomized to initiate medications for the treatment for AUD in the ED in addition to receiving a brief intervention and referral to ongoing treatment, which all participants will receive.

The secondary objective of this study is to evaluate the difference in reduction of heavy drinking days between the two ED treatment models during the 30 days post ED visit.

DETAILED DESCRIPTION:
The proposed study will evaluate a comprehensive ED-based intervention for moderate to severe AUD combining SBIRT with ED-initiated MAUD. It is an extension and a novel application of a highly effective ED intervention model that has been successfully developed and broadly disseminated for other conditions, such as diabetes, hypertension and more recently opioid use disorder. No prospective randomized controlled trials of ED-initiated medications for the treatment of AUD, with or without psychosocial interventions, have been published to date. If found efficacious this novel intervention model has a potential to increase AUD treatment participation rates among individuals with AUD who frequently receive care in the ED. The proposed study will evaluate two ED-based interventions that have a potential to be broadly disseminated to narrow the gap between treatment need and treatment access.

Study participants will be identified through targeted screening for DSM-5 criteria for moderate to severe AUD and the study inclusion/exclusion criteria. Therefore, the Screening component of the SBIRT intervention in the proposed RCT will be conducted before eligible ED patients who are interested in study participation are consented and randomized. This study will compare outcomes among individuals who are initiated on MAUD treatment in the ED, including AUD treatment with naltrexone, with ancillary support of gabapentin to assist with withdrawal symptoms.

Hypothesis 1: The rates of AUD treatment engagement will be higher among patients receiving SBIRT+ED-MAUD.

Hypothesis 2: Those randomized to SBIRT+ED-MAUD will have greater reductions of heavy drinking days.

This study is not designed to change the FDA labeling of gabapentin.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 80 years in age
2. Diagnosed with moderate to severe Alcohol Use Disorder
3. Stated willingness and ability to comply with all study procedures and availability for the duration of the study
4. Reproductive aged females will have a negative pregnancy test within the past 24 hours and agree to use of highly effective family planning during study participation period
5. Able to speak English sufficiently to understand study procedures and provide written informed consent to participate in the study.
6. Clinical Alcohol Withdrawal Scale (CIWA-Ar) ≥ 4.

Exclusion Criteria:

1. A current diagnosis of OUD, self-reported past 7 day opioid or opioid pain medication use, or a positive urine opioid screen (opiates, methadone, buprenorphine, oxycodone, hydrocodone, tramadol and fentanyl)
2. Current prescription of opioid pain medications, or anticipated need for opioid pain medications during the study period (i.e. planned surgery)
3. History of complicated alcohol withdrawal
4. Condition that precludes interview (i.e., life threatening injury/illness)
5. Inability to consent due to cognitive impairment
6. Awaiting an acute psychiatric evaluation for psychosis or suicidal ideation
7. In police custody
8. Unable to provide contact information
9. Previously enrolled in this study or currently enrolled in another study for which they are currently receiving study medications or active ongoing intervention
10. Any contraindication to naltrexone or gabapentin, including known allergy, renal failure, acute hepatitis, hepatic failure,1 or severe lung disease or other chronic conditions such as chronic obstructive pulmonary disease (COPD).
11. Creatine Clearance <60 mL/min within past 72 hours.
12. Currently pregnant or breast feeding
13. Requiring hospitalization at the time of the index visit
14. Past week treatment with medications for the treatment of alcohol use disorder
15. Taking gabapentin or naltrexone for any reason
16. Appearing unable or unwilling to comply with discharge instructions or complete follow-up
17. Current residence outside of the state of Connecticut

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Participation in AUD Treatment on Day 30 post-randomization | 30 days post enrollment
  The proportions of participants participating in AUD treatment on day 30 post enrollment in SBIRT and SBIRT+EDMAUD groups.

SECONDARY OUTCOMES:
Days of heavy alcohol drinking | 30 days post ED visit
  The number of heavy alcohol drinking days during the 30 days prior and during 30 days post the ED index visit. This outcome will be based on self-report using the timeline follow-back (TLFB) method. A day of heavy alcohol drinking is defined by the NIAAA criteria as: for men, consuming more than 4 drinks on any day; for women, consuming more than 3 drinks on any day.
AUD Treatment Linkage | up to 7 days post ED visit
  The proportion of participants that initiate AUD treatment within 7 days post ED visit with providers to which they were referred during the ED visit
Alcohol craving | up to 7 days post enrollment
  Daily intensity of alcohol craving measured on a visual analog scale of 0 to 100.
Alcohol withdrawal symptoms | up to 7 days post enrollment
  Daily intensity of alcohol withdrawal measured on a visual analog scale of 0 to 100.
Daily naltrexone medication adherence | up to 7 days post enrollment
  Number of oral naltrexone doses taken in the past 24 hours for 7 days post enrollment of those initiated on oral naltrexone in the SBIRT+ED- MAUD arm.
Daily gabapentin medication adherence | up to 7 days post enrollment
  Number of gabapentin doses taken in the past 24 hours of those in the SBIRT+ED- MAUD arm.
Treatment linkage | 7 days
  • Proportion of patients in each of the two study arms initiating outpatient AUD treatment within 7 days post the ED visit with providers to which they were referred during the ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Hawk, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available through NIAAA Data Archive